CLINICAL TRIAL: NCT01308567
Title: Randomized, Open Label, Multi-Center Study Comparing Cabazitaxel at 25 mg/m^2 and at 20 mg/m^2 in Combination With Prednisone Every 3 Weeks to Docetaxel in Combination With Prednisone in Patients With Metastatic Castration Resistant Prostate Cancer Not Pretreated With Chemotherapy
Brief Title: Cabazitaxel Versus Docetaxel Both With Prednisone in Patients With Metastatic Castration Resistant Prostate Cancer
Acronym: FIRSTANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11784; 2010-022064-12 (EudraCT Number); U1111-1117-8356 (Other: UTN)
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cabazitaxel 25 mg/m^2 (Experimental): Cabazitaxel 25 mg/m^2 intravenous (IV) infusion on Day 1 of each 21-day cycle in combination with Prednisone 10 mg orally, once daily until disease progression (DP), unacceptable toxicity or participant's refusal.
  Interventions: Drug: Cabazitaxel (XRP6258); Drug: Prednisone
- Cabazitaxel 20 mg/m^2 (Experimental): Cabazitaxel 20 mg/m^2 IV infusion on Day 1 of each 21 -day cycle in combination with Prednisone 10 mg orally, once daily until DP, unacceptable toxicity or participant's refusal.
  Interventions: Drug: Cabazitaxel (XRP6258); Drug: Prednisone
- Docetaxel 75 mg/m^2 (Active Comparator): Docetaxel (TXT) 75 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with Prednisone 10 mg orally, once daily until DP, unacceptable toxicity or participant's refusal.
  Interventions: Drug: Docetaxel (XRP6976); Drug: Prednisone

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form: Solution for injection; Route of administration: Intravenous
  Arms: Cabazitaxel 20 mg/m^2; Cabazitaxel 25 mg/m^2
Drug: Docetaxel (XRP6976) — Pharmaceutical form: Solution for injection'; Route of administration: Intravenous
  Arms: Docetaxel 75 mg/m^2
Drug: Prednisone — Pharmaceutical form: Tablet; Route of administration: Oral

SUMMARY:
Primary Objective:

* To demonstrate the superiority of cabazitaxel plus prednisone at 25 mg/m^2 (Arm A) or 20 mg/m^2 (Arm B) versus docetaxel plus prednisone (Arm C) in term of overall survival (OS) in participants with metastatic castration resistant prostate cancer (mCRPC) and not previously treated with chemotherapy.

Secondary Objectives:

* To evaluate safety in the 3 treatment arms.
* To compare efficacy of cabazitaxel at 20 mg/m^2 and 25 mg/m^2 to docetaxel for:

  * Progression Free Survival (PFS) (RECIST 1.1)
  * Tumor progression free survival (RECIST 1.1)
  * Tumor response in participants with measurable disease (RECIST 1.1),
  * PSA response
  * PSA-Progression free survival (PSA-PFS).
  * Pain response in participants with stable pain at baseline
  * Pain progression free survival
  * Time to occurrence of any skeletal related events (SRE)
* To compare Health-Related Quality of Life (HRQL).
* To assess the pharmacokinetics and pharmacogenomics of cabazitaxel.

DETAILED DESCRIPTION:
Participants were treated until progressive disease, unacceptable toxicity, or participant's refusal of further study treatment. All participants were followed when on study treatment and after completion of study treatment during follow up period until death or the study cutoff date, whichever comes first.

ELIGIBILITY:
Inclusion criteria :

* I 01. Histologically- or cytologically-confirmed prostate adenocarcinoma.
* I 02. Metastatic disease.
* I 03. Progressive disease while receiving hormonal therapy or after surgical castration.
* I 04. Effective castration (serum testosterone levels ≤0.50 ng/mL) by orchiectomy and/or luteinizing hormone-releasing hormone (LHRH) agonists or antagonist with or without anti-androgens.

Exclusion criteria:

* E 01. Prior chemotherapy for prostate cancer,
* E 02. Less than 28 days elapsed from prior treatment with estramustine, radiotherapy or surgery to the time of randomization. Participants on biphosphonates prior to study entry.
* E 03. Prior isotope therapy, whole pelvic radiotherapy, or radiotherapy to >30% of bone marrow.
* E 04. Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of grade >1(National Cancer Institute Common Terminology Criteria [NCI CTCAE] v4.03) at the time of randomization.
* E 05. Less than 18 years (or country's legal age of majority if the legal age is >18 years).
* E 06. Eastern Cooperative Oncology Group (ECOG) performance status >2.
* E 07. History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* E 08. Prior malignancy.
* E 09. Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.
* E 10. Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack.
* E 11. Any of the following within 3 months prior to randomization: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
* E 12. Acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
* E 13. Any severe acute or chronic medical condition which could impair the ability of the participant to participate to the study or interfere with interpretation of study results, or participants unable to comply with the study procedures.
* E 14. Absence of signed and dated Institutional Review Board (IRB)-approved participant informed consent form prior to enrollment into the study.
* E 15. Participants with reproductive potential who did not agree to use accepted and effective method of contraception during the study treatment period.
* E 16. History of hypersensitivity to docetaxel, or polysorbate 80.
* E 17. Inadequate organ and bone marrow function
* E 18. Contraindications to the use of corticosteroid treatment.
* E 19. Symptomatic peripheral neuropathy grade >2 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] v.4.03).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (167):
- United States (32):
  - Investigational Site Number 840004, Muscle Shoals, Alabama
  - Investigational Site Number 840009, Anaheim, California
  - Investigational Site Number 840014, Bakersfield, California
  - Investigational Site Number 840030, Sacramento, California
  - Investigational Site Number 840003, San Bernardino, California
  - Investigational Site Number 840012, San Francisco, California
  - Investigational Site Number 840019, Denver, Colorado
  - Investigational Site Number 840013, Boca Raton, Florida
  - Investigational Site Number 840035, Jacksonville, Florida
  - Investigational Site Number 840001, Port Saint Lucie, Florida
  - Investigational Site Number 840015, Decatur, Illinois
  - Investigational Site Number 840018, Wichita, Kansas
  - Investigational Site Number 840010, Paducah, Kentucky
  - Investigational Site Number 840008, New Orleans, Louisiana
  - Investigational Site Number 840006, Rockville, Maryland
  - Investigational Site Number 840238, Boston, Massachusetts
  - Investigational Site Number 840138, Boston, Massachusetts
  - Investigational Site Number 840038, Brookline, Massachusetts
  - Investigational Site Number 840005, Detroit, Michigan
  - Investigational Site Number 840021, Saint Louis Park, Minnesota
  - Investigational Site Number 840016, Kansas City, Missouri
  - Investigational Site Number 840020, Lincoln, Nebraska
  - Investigational Site Number 840017, East Orange, New Jersey
  - Investigational Site Number 840033, Albuquerque, New Mexico
  - Investigational Site Number 840036, Raleigh, North Carolina
  - Investigational Site Number 840011, Washington, North Carolina
  - Investigational Site Number 840026, Akron, Ohio
  - Investigational Site Number 840023, Cleveland, Ohio
  - Investigational Site Number 840032, Dunmore, Pennsylvania
  - Investigational Site Number 840007, Pawtucket, Rhode Island
  - Investigational Site Number 840037, Myrtle Beach, South Carolina
  - Investigational Site Number 840028, Chattanooga, Tennessee
- Australia (12):
  - Investigational Site Number 036016, Bankstown
  - Investigational Site Number 036008, Camperdown
  - Investigational Site Number 036015, Coffs Harbour
  - Investigational Site Number 036001, Concord
  - Investigational Site Number 036017, Fitzroy
  - Investigational Site Number 036003, Herston
  - Investigational Site Number 036010, Hornsby
  - Investigational Site Number 036012, Kurralta Park
  - Investigational Site Number 036002, Parkville
  - Investigational Site Number 036009, South Brisbane
  - Investigational Site Number 036011, Subiaco
  - Investigational Site Number 036013, Wodonga
- Belarus (3):
  - Investigational Site Number 112001, Minsk
  - Investigational Site Number 112002, Minsk
  - Investigational Site Number 112004, Vitebsk
- Brazil (7):
  - Investigational Site Number 076006, Passo Fundo
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076002, Porto Alegre
  - Investigational Site Number 076004, Rio de Janeiro
  - Investigational Site Number 076009, São José do Rio Preto
  - Investigational Site Number 076005, São Paulo
  - Investigational Site Number 076003, Uberlândia
- Canada (6):
  - Investigational Site Number 124002, London
  - Investigational Site Number 124007, Mississauga
  - Investigational Site Number 124005, Moncton
  - Investigational Site Number 124003, Montreal
  - Investigational Site Number 124004, Québec
  - Investigational Site Number 124006, Toronto
- China (4):
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156002, Shanghai
  - Investigational Site Number 156003, Shanghai
  - Investigational Site Number 156004, Shanghai
- Czechia (4):
  - Investigational Site Number 203002, Brno
  - Investigational Site Number 203003, Nový Jičín
  - Investigational Site Number 203001, Olomouc
  - Investigational Site Number 203004, Prague
- Denmark (4):
  - Investigational Site Number 208004, Aalborg
  - Investigational Site Number 208002, Herlev
  - Investigational Site Number 208001, København Ø
  - Investigational Site Number 208003, Odense C
- Finland (3):
  - Investigational Site Number 246002, Helsinki
  - Investigational Site Number 246001, Kuopio
  - Investigational Site Number 246003, Turku
- France (10):
  - Investigational Site Number 250010, Besançon
  - Investigational Site Number 250002, Bordeaux
  - Investigational Site Number 250006, Caen
  - Investigational Site Number 250005, Lyon
  - Investigational Site Number 250003, Paris
  - Investigational Site Number 250004, Paris
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250007, Poitiers
  - Investigational Site Number 250008, Suresnes
  - Investigational Site Number 250009, Villejuif
- Germany (6):
  - Investigational Site Number 276003, Aachen
  - Investigational Site Number 276005, Berlin
  - Investigational Site Number 276001, Düsseldorf
  - Investigational Site Number 276004, Erlangen
  - Investigational Site Number 276002, Homburg
  - Investigational Site Number 276006, München
- Israel (3):
  - Investigational Site Number 376004, Kfar Saba
  - Investigational Site Number 376003, Petah Tikva
  - Investigational Site Number 376002, Tel Aviv
- Italy (5):
  - Investigational Site Number 380001, Arezzo
  - Investigational Site Number 380004, Bari
  - Investigational Site Number 380003, Orbassano
  - Investigational Site Number 380005, Roma
  - Investigational Site Number 380002, Trento
- Japan (6):
  - Investigational Site Number 392001, Bunkyō City
  - Investigational Site Number 392003, Chiba
  - Investigational Site Number 392006, Kashiwa-Shi
  - Investigational Site Number 392005, Kōtoku
  - Investigational Site Number 392004, Osaka
  - Investigational Site Number 392002, Osaka Sayama-Shi
- Mexico (8):
  - Investigational Site Number 484007, Acapulco
  - Investigational Site Number 484008, Aguascalientes
  - Investigational Site Number 484003, D.F.
  - Investigational Site Number 484004, Guadalajara
  - Investigational Site Number 484009, Mérida
  - Investigational Site Number 484005, Querétaro
  - Investigational Site Number 484002, San Luis Potosí City
  - Investigational Site Number 484006, Zapopan
- Peru (4):
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604002, Lima
- Poland (5):
  - Investigational Site Number 616002, Bydgoszcz
  - Investigational Site Number 616001, Gdansk
  - Investigational Site Number 616003, Kościerzyna
  - Investigational Site Number 616005, Lodz
  - Investigational Site Number 616004, Poznan
- Portugal (5):
  - Investigational Site Number 620003, Coimbra
  - Investigational Site Number 620005, Lisbon
  - Investigational Site Number 620004, Lisbon
  - Investigational Site Number 620001, Porto
  - Investigational Site Number 620002, Porto
- Romania (6):
  - Investigational Site Number 642004, Baia Mare
  - Investigational Site Number 642005, Bucharest
  - Investigational Site Number 642008, Bucharest
  - Investigational Site Number 642002, Cluj-Napoca
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642007, Hunedoara
- Russia (8):
  - Investigational Site Number 643008, Moscow
  - Investigational Site Number 643003, Omsk
  - Investigational Site Number 643002, Pyatigorsk
  - Investigational Site Number 643007, Ryazan
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643001, Tomsk
  - Investigational Site Number 643006, Yaroslavl
  - Investigational Site Number 643004, Yekaterinburg
- Spain (7):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724007, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724003, L'Hospitalet de Llobregat
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724006, Santiago de Compostela
- Sweden (3):
  - Investigational Site Number 752003, Malmo
  - Investigational Site Number 752002, Stockholm
  - Investigational Site Number 752001, Uppsala
- Taiwan (4):
  - Investigational Site Number 158004, Kaohsiung City
  - Investigational Site Number 158002, Taichung
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158003, Taoyuan District
- Turkey (Türkiye) (2):
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792001, Istanbul
- Ukraine (10):
  - Investigational Site Number 804009, Cherkasy
  - Investigational Site Number 804004, Dnipropetrovsk
  - Investigational Site Number 804010, Donetsk
  - Investigational Site Number 804006, Ivano-Frankivsk
  - Investigational Site Number 804003, Kharkiv
  - Investigational Site Number 804002, Kyiv
  - Investigational Site Number 804001, Kyiv
  - Investigational Site Number 804007, Lutsk
  - Investigational Site Number 804005, Uzhhorod
  - Investigational Site Number 804008, Zaporizhzhya

REFERENCES:
- [Derived] Carrot A, Oudard S, Colomban O, Fizazi K, Maillet D, Sartor O, Freyer G, You B. Prognostic Value of the Modeled Prostate-Specific Antigen KELIM Confirmation in Metastatic Castration-Resistant Prostate Cancer Treated With Taxanes in FIRSTANA. JCO Clin Cancer Inform. 2024 Feb;8:e2300208. doi: 10.1200/CCI.23.00208. PMID 38364191
- [Derived] Thiery-Vuillemin A, Fizazi K, Sartor O, Oudard S, Bury D, Thangavelu K, Ozatilgan A, Poole EM, Eisenberger M, de Bono J. An analysis of health-related quality of life in the phase III PROSELICA and FIRSTANA studies assessing cabazitaxel in patients with metastatic castration-resistant prostate cancer. ESMO Open. 2021 Apr;6(2):100089. doi: 10.1016/j.esmoop.2021.100089. Epub 2021 Mar 16. PMID 33740734
- [Derived] Mehra N, Dolling D, Sumanasuriya S, Christova R, Pope L, Carreira S, Seed G, Yuan W, Goodall J, Hall E, Flohr P, Boysen G, Bianchini D, Sartor O, Eisenberger MA, Fizazi K, Oudard S, Chadjaa M, Mace S, de Bono JS. Plasma Cell-free DNA Concentration and Outcomes from Taxane Therapy in Metastatic Castration-resistant Prostate Cancer from Two Phase III Trials (FIRSTANA and PROSELICA). Eur Urol. 2018 Sep;74(3):283-291. doi: 10.1016/j.eururo.2018.02.013. Epub 2018 Feb 28. PMID 29500065
- [Derived] Oudard S, Fizazi K, Sengelov L, Daugaard G, Saad F, Hansen S, Hjalm-Eriksson M, Jassem J, Thiery-Vuillemin A, Caffo O, Castellano D, Mainwaring PN, Bernard J, Shen L, Chadjaa M, Sartor O. Cabazitaxel Versus Docetaxel As First-Line Therapy for Patients With Metastatic Castration-Resistant Prostate Cancer: A Randomized Phase III Trial-FIRSTANA. J Clin Oncol. 2017 Oct 1;35(28):3189-3197. doi: 10.1200/JCO.2016.72.1068. Epub 2017 Jul 28. PMID 28753384
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- [Derived] Winquist E, Rodrigues G. Open clinical uro-oncology trials in Canada. Can J Urol. 2012 Dec;19(6):6587-91. No abstract available. PMID 23228299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 159 centers in 25 countries. A total of 1510 participants were screened between 17 May 2011 and 09 September 2015 of whom 1168 participants were randomized and 342 were considered as screen failures.
Pre-assignment Details: A total of 1168 participants randomized in this study. Of these, 21 participants randomized but not treated. These participants were included in intent-to-treat (ITT) population, not in safety population. "Study cut-off date" for outcome measures was up to "primary completion date" (PCD) only. After PCD, only adverse event (AE) data was updated.
Groups:
- Docetaxel 75 mg/m^2: Docetaxel (TXT) 75 mg/m^2 intravenous (IV) infusion on Day 1 of each 21-day cycle in combination with Prednisone 10 mg orally, once daily until disease progression (DP), unacceptable toxicity or participant's refusal.
- Cabazitaxel 20 mg/m^2: Cabazitaxel 20 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with Prednisone 10 mg orally, once daily until DP, unacceptable toxicity or participant's refusal.
- Cabazitaxel 25 mg/m^2: Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with Prednisone 10 mg orally, once daily until DP, unacceptable toxicity or participant's refusal.
Period: Overall Study
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Started | 391 (Randomized) | 389 (Randomized) | 388 (Randomized)
Treated | 388 (For 1 participant, actual treatment received was Cabazitaxel 25 mg/m^2.) | 382 (For 15 participants, actual treatment received was Cabazitaxel 25 mg/m^2.) | 377 (For 2 participants, actual treatment received was Cabazitaxel 20 mg/m^2.)
Completed | 389 (Completed participants included those who withdrew treatment consent but were followed for survival.) | 385 (Completed participants included those who withdrew treatment consent but were followed for survival.) | 384 (Completed participants included those who withdrew treatment consent but were followed for survival.)
Not Completed | 2 | 4 | 4
Not completed — Lost to Follow-up | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2 | Total
Number analyzed (Participants) | 391 | 389 | 388 | 1168
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 123 | 128 | 125 | 376
  65-74 years | 181 | 187 | 182 | 550
  ≥75 years | 87 | 74 | 81 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 391 | 389 | 388 | 1168

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date participant was known to be alive, or at the cut-off date if the participant's last contact was after the cut-off date. The study cut-off date for the final analysis of OS was the date when the 774th death had been observed. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline up to death or study cut-off date, whichever was earlier (maximum duration: 51 months )
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 24.3 [22.18 to 27.60] | 24.5 [21.75 to 27.20] | 25.2 [22.90 to 26.97]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; Hazard ratio was estimated using a Cox Proportional Hazards regression model. The Cox proportional hazard model was adjusted by Eastern Cooperative Oncology Group performance status (ECOG PS) score at baseline, measurable disease at baseline, and region with commercial availability of cabazitaxel at the time of randomization; Test type: Superiority or Other; p = 0.7574, Log Rank — P-value from two-sided stratified log-rank test, stratified for ECOG PS score at baseline, measurable disease at baseline and region with commercial availability of cabazitaxel at time of randomization. Threshold for statistical significance = 0.0479; Hazard Ratio (HR) = 0.975, 95% CI 2-sided [0.819 to 1.16] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; Hazard ratio was estimated using a Cox Proportional Hazards regression model. The Cox proportional hazard model was adjusted by ECOG PS score at baseline, measurable disease at baseline, and region with commercial availability of cabazitaxel at the time of randomization; Test type: Superiority or Other; p = 0.9967, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.009, 95% CI 2-sided [0.85 to 1.197] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: time interval between date of randomization to date of first occurrence of any of following events: tumor progression according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1; Prostate Specific Antigen (PSA) progression; pain progression or death due to any cause. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline up to tumor progression, PSA progression, pain progression or death (maximum duration: 51 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 5.3 [4.86 to 5.78] | 4.4 [3.91 to 5.09] | 5.1 [4.60 to 5.72]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.989, 95% CI 2-sided [0.849 to 1.152] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.063, 95% CI 2-sided [0.913 to 1.236] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

3. Secondary Outcome: Time to Tumor Progression Free Survival
Description: Time to tumor progression free survival was defined as the time interval between randomization and the date of first occurrence of tumor progression (assessed using RECIST version 1.1) or death, whichever was earlier. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline up to tumor progression or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 51 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 12.1 [11.30 to 13.77] | 13.4 [11.37 to 14.75] | 13.1 [11.66 to 14.32]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.958, 95% CI 2-sided [0.785 to 1.17] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.916, 95% CI 2-sided [0.75 to 1.118] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

4. Secondary Outcome: Percentage of Participants With Overall Objective Tumor Response
Description: Overall objective tumor response was defined as having a partial response (PR) or complete response (CR) according to the RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to DP or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 51 months)
Population: Analysis was performed on ITT population. Number of participants analyzed=participants with measurable disease at baseline and at least one valid post-baseline value analyzed for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 175 | 188 | 173
percentage of participants | 30.9 [24.0 to 37.7] | 32.4 [25.8 to 39.1] | 41.6 [34.3 to 49.0]

5. Secondary Outcome: Time to Prostate Serum Antigen Progression Free Survival (PSA-PFS)
Description: Time to PSA-PFS: time interval between date of randomization & first occurrence of PSA progression/ death, whichever was earlier. PSA progression:1) In PSA responders(≥50% decline from baseline PSA of ≥10 ng/mL):increase of ≥25%(at least 2 ng/mL)over nadir value, confirmed by second PSA value at least 3 weeks later;2)In PSA non-responders(not achieved ≥50% decline from baseline PSA ≥10 ng/mL):increase of ≥25% (at least 2 ng/mL) over baseline value, confirmed by second PSA value at least 3 weeks later;3)In participants not eligible for PSA response(baseline PSA <10 ng/mL):(a)in participants with baseline PSA>0 ng/mL&<10 ng/mL: increase in PSA by 25% (at least 2 ng/mL) above baseline level, confirmed by second PSA value at least 3weeks apart;(b)in participants with baseline value=0ng/mL: a post baseline PSA value ≥2ng/mL.Early rise in PSA only indicated progression if it was associated with another sign of DP or if it continued beyond 12 weeks. Analysis performed by Kaplan-Meier method.
Time Frame: Baseline up to PSA progression or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 51 months)
Population: Analysis was performed on ITT population which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 8.3 [7.66 to 9.20] | 8.2 [7.43 to 8.90] | 9.2 [8.44 to 9.92]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.8 to 1.123] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.886 to 1.238] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

6. Secondary Outcome: Percentage of Participants With PSA Response
Description: PSA response was defined as ≥50% decrease from baseline in serum PSA levels, confirmed by a second PSA value at least 3 weeks later in participants with baseline PSA value ≥10 ng/mL.
Time Frame: as for outcome 5
Population: Analysis was performed on ITT population. Number of participants analyzed=participants with PSA value ≥10 ng/mL at baseline and at least one valid post-baseline value for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 354 | 346 | 342
percentage of participants | 68.4 [63.5 to 73.2] | 60.7 [55.5 to 65.8] | 68.7 [63.8 to 73.6]

7. Secondary Outcome: Time to Pain Progression Free Survival (Pain PFS)
Description: Time to pain PFS was defined as the time interval between date of randomization and the date of the first occurrence of pain progression or death, whichever was earlier. Pain progression was defined as an increase of ≥1 point in the median present pain intensity (PPI) score from the nadir confirmed by a second assessment at least 3 weeks later or ≥25 % increase in the mean analgesic score from baseline, due to cancer related pain confirmed by a second assessment at least 3 weeks later or requirement for local palliative radiotherapy. PPI was rated by participant in a diary using a scale of 0=no pain, 1=mild, 2=discomforting, 3=distressing, 4=horrible 5=excruciating. Analgesic use was recorded by the participant in a diary. Analgesic score was calculated from the analgesic use data based on a table of analgesic medications, with non-narcotic medications assigned a value of 1 point and narcotic medications assigned a value of 4 points. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until disease progression, death or study cut-off date (maximum duration: 51 months)
Population: Analysis was performed on ITT population which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 10.1 [8.28 to 11.76] | 8.0 [6.90 to 9.66] | 7.3 [6.44 to 9.30]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.189, 95% CI 2-sided [0.986 to 1.434] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.189, 95% CI 2-sided [0.985 to 1.435] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

8. Secondary Outcome: Percentage of Participants With Pain Response
Description: Pain response was defined as either a ≥2-point decrease from baseline median PPI score without increase in analgesic score, or a ≥50% decrease in analgesic use from baseline mean analgesic score (only in participants with baseline mean analgesic score≥10) without increase in the pain. Either criterion was maintained for 2 consecutive evaluations at least 3 weeks apart. PPI was rated by participant in a diary using a scale of 0=no pain, 1=mild, 2=discomforting, 3=distressing, 4=horrible 5=excruciating. Analgesic use was recorded by the participant in a diary. Analgesic score was calculated from the analgesic use data based on a table of analgesic medications, with non-narcotic medications assigned a value of 1 point and narcotic medications assigned a value of 4 points.
Time Frame: Baseline until pain progression, death or study cut-off date (maximum duration: 51 months)
Population: Analysis was performed on ITT population. Number of participants analyzed=participants with pain score with median PPI >= 2 and/or mean analgesic score >= 10 points at baseline and at least one valid post-baseline value for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 81 | 99 | 104
percentage of participants | 40.7 [30.0 to 51.4] | 42.4 [32.7 to 52.2] | 39.4 [30.0 to 48.8]

9. Secondary Outcome: Skeletal Related Events (SRE) Free Survival
Description: SRE free survival was defined as the time interval between the date of randomization and the date of the occurrence of the first event defining a SRE or death due to any cause, whichever was earlier. SRE were assessed by clinical evaluation. Occurrence of SRE was defined as: pathological fracture(s) and/or spinal cord compression; need for bone irradiation, including radioisotopes or bone surgery; and change of antineoplastic therapy (including introduction of bisphosphonates or denosumab in the setting of increased pain) to treat bone pain. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until occurrence of first SRE or death (maximum duration: 51 months)
Population: Analysis was performed on ITT population which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 391 | 389 | 388
months | 19.0 [15.24 to 22.44] | 19.2 [15.21 to 24.61] | 17.1 [14.59 to 20.50]
Statistical Analysis 1: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.121, 95% CI 2-sided [0.886 to 1.417] — Cabazitaxel 25 mg/m^2 vs Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Docetaxel 75 mg/m^2 vs Cabazitaxel 20 mg/m^2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.014, 95% CI 2-sided [0.798 to 1.288] — Cabazitaxel 20 mg/m^2 vs Docetaxel 75 mg/m^2

10. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Total Score as a Measure of Health Related Quality of Life (HRQoL)
Description: FACT-P was a 39-item participant rated questionnaire that measures the concerns of participants with prostate cancer. It consisted of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). FACT-P total score was the sum of all 5 subscale scores. It ranged from 0 to156 with higher score indicated better quality of life with fewer symptoms.
Time Frame: Baseline, Day 1 of each cycle 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16 (each cycle 21-day); post-treatment follow up 1, 2, 3, 4, 5, 6 (each up to 12 weeks)
Population: Analysis was performed on FACT-P population that included all participants with evaluable individual FACT-P subscale score at baseline and post-baseline on at least 1 of the subscale domains. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 375 | 370 | 361
units on a scale
  Change at Cycle 1: number analyzed (Participants) | 333 | 323 | 321
  Change at Cycle 1 | 4.17 [1.3 to 7.05] | 7.66 [4.79 to 10.53] | 6.93 [3.97 to 9.88]
  Change at Cycle 2: number analyzed (Participants) | 339 | 339 | 323
  Change at Cycle 2 | 5.33 [2.46 to 8.2] | 7.15 [4.28 to 10.01] | 5.28 [2.32 to 8.24]
  Change at Cycle 3: number analyzed (Participants) | 330 | 332 | 316
  Change at Cycle 3 | 4.94 [2.06 to 7.82] | 6.79 [3.93 to 9.66] | 4.61 [1.64 to 7.58]
  Change at Cycle 4: number analyzed (Participants) | 316 | 323 | 302
  Change at Cycle 4 | 4.07 [1.17 to 6.96] | 5.22 [2.35 to 8.09] | 4.01 [1.03 to 6.99]
  Change at Cycle 5: number analyzed (Participants) | 293 | 290 | 283
  Change at Cycle 5 | 4.36 [1.44 to 7.27] | 5.16 [2.26 to 8.06] | 4.09 [1.09 to 7.08]
  Change at Cycle 6: number analyzed (Participants) | 272 | 267 | 262
  Change at Cycle 6 | 3.46 [0.53 to 6.39] | 3.8 [0.88 to 6.73] | 3.37 [0.35 to 6.39]
  Change at Cycle 7: number analyzed (Participants) | 244 | 246 | 241
  Change at Cycle 7 | 3.16 [0.2 to 6.12] | 3.66 [0.71 to 6.61] | 3.42 [0.38 to 6.45]
  Change at Cycle 8: number analyzed (Participants) | 228 | 222 | 225
  Change at Cycle 8 | 2.61 [-0.37 to 5.59] | 2.71 [-0.27 to 5.68] | 1.67 [-1.39 to 4.73]
  Change at Cycle 9: number analyzed (Participants) | 174 | 196 | 190
  Change at Cycle 9 | 2.2 [-0.87 to 5.27] | 2.67 [-0.35 to 5.68] | 1.89 [-1.22 to 5.01]
  Change at Cycle 10: number analyzed (Participants) | 149 | 164 | 166
  Change at Cycle 10 | 2.08 [-1.05 to 5.21] | 2.09 [-0.99 to 5.18] | 1.84 [-1.32 to 5]
  Change at Cycle 11: number analyzed (Participants) | 101 | 115 | 111
  Change at Cycle 11 | 0.15 [-3.18 to 3.47] | 3.35 [0.1 to 6.6] | 2.68 [-0.67 to 6.02]
  Change at Cycle 12: number analyzed (Participants) | 83 | 98 | 98
  Change at Cycle 12 | 0.52 [-2.94 to 3.97] | 3.95 [0.61 to 7.29] | 0.63 [-2.78 to 4.05]
  Change at Cycle 13: number analyzed (Participants) | 58 | 85 | 80
  Change at Cycle 13 | 1.79 [-1.94 to 5.53] | 2.48 [-0.95 to 5.91] | 0.55 [-3 to 4.09]
  Change at Cycle 14: number analyzed (Participants) | 55 | 78 | 71
  Change at Cycle 14 | -1.78 [-5.56 to 2] | 2.2 [-1.29 to 5.69] | -0.42 [-4.06 to 3.21]
  Change at Cycle 15: number analyzed (Participants) | 44 | 71 | 63
  Change at Cycle 15 | -3.49 [-7.5 to 0.51] | 1.74 [-1.82 to 5.3] | 1.22 [-2.51 to 4.95]
  Change at Cycle 16: number analyzed (Participants) | 42 | 58 | 58
  Change at Cycle 16 | -3.83 [-7.89 to 0.23] | 1.62 [-2.11 to 5.35] | 0.5 [-3.3 to 4.3]
  Change at Follow-up 1: number analyzed (Participants) | 176 | 185 | 175
  Change at Follow-up 1 | -1.08 [-4.15 to 1.99] | -1.45 [-4.48 to 1.59] | -1.82 [-4.97 to 1.32]
  Change at Follow-up 2: number analyzed (Participants) | 145 | 129 | 133
  Change at Follow-up 2 | -0.02 [-3.16 to 3.13] | -1.98 [-5.17 to 1.21] | -1.78 [-5.04 to 1.47]
  Change at Follow-up 3: number analyzed (Participants) | 110 | 103 | 101
  Change at Follow-up 3 | -0.55 [-3.83 to 2.74] | -2.16 [-5.47 to 1.14] | -2.68 [-6.08 to 0.72]
  Change at Follow-up 4: number analyzed (Participants) | 87 | 73 | 81
  Change at Follow-up 4 | -1.19 [-4.61 to 2.23] | -3.64 [-7.18 to -0.1] | -1.7 [-5.25 to 1.84]
  Change at Follow-up 5: number analyzed (Participants) | 72 | 63 | 76
  Change at Follow-up 5 | -2.05 [-5.61 to 1.51] | -6.73 [-10.39 to -3.06] | -0.6 [-4.18 to 2.99]
  Change at Follow-up 6: number analyzed (Participants) | 58 | 46 | 57
  Change at Follow-up 6 | -1.17 [-4.92 to 2.58] | -5.36 [-9.32 to -1.4] | -4.05 [-7.87 to -0.23]

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P):Trial Outcome Index (TOI) as a Measure of HRQoL
Description: FACT-P was a 39-item participant rated questionnaire that measures the concerns of participants with prostate cancer. It consisted of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). Physical well being, functional well being, and prostate-specific concerns sub-scales of the FACT-P questionnaire were combined to calculate TOI. Total TOI score ranges from 0 to 104, with higher scores representing a better quality of life with fewer symptoms.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 376 | 371 | 361
units on a scale
  Change at Cycle 1: number analyzed (Participants) | 331 | 324 | 318
  Change at Cycle 1 | 3.31 [1.05 to 5.58] | 6.09 [3.83 to 8.35] | 5.76 [3.43 to 8.09]
  Change at Cycle 2: number analyzed (Participants) | 334 | 337 | 318
  Change at Cycle 2 | 4.37 [2.1 to 6.64] | 5.96 [3.7 to 8.21] | 4.26 [1.92 to 6.59]
  Change at Cycle 3: number analyzed (Participants) | 325 | 332 | 314
  Change at Cycle 3 | 4.31 [2.04 to 6.58] | 5.28 [3.02 to 7.53] | 3.65 [1.31 to 5.99]
  Change at Cycle 4: number analyzed (Participants) | 313 | 321 | 301
  Change at Cycle 4 | 3.39 [1.11 to 5.67] | 4.1 [1.83 to 6.36] | 3.2 [0.85 to 5.55]
  Change at Cycle 5: number analyzed (Participants) | 289 | 285 | 282
  Change at Cycle 5 | 3.41 [1.11 to 5.7] | 4.05 [1.76 to 6.34] | 3.1 [0.74 to 5.46]
  Change at Cycle 6: number analyzed (Participants) | 270 | 264 | 260
  Change at Cycle 6 | 2.76 [0.45 to 5.07] | 3.15 [0.85 to 5.46] | 2.88 [0.5 to 5.26]
  Change at Cycle 7: number analyzed (Participants) | 239 | 241 | 240
  Change at Cycle 7 | 2.29 [-0.05 to 4.62] | 3.14 [0.81 to 5.47] | 2.94 [0.54 to 5.34]
  Change at Cycle 8: number analyzed (Participants) | 223 | 220 | 222
  Change at Cycle 8 | 1.67 [-0.69 to 4.02] | 2.26 [-0.09 to 4.61] | 1.49 [-0.92 to 3.91]
  Change at Cycle 9: number analyzed (Participants) | 174 | 192 | 189
  Change at Cycle 9 | 1.75 [-0.67 to 4.18] | 2.15 [-0.24 to 4.53] | 1.73 [-0.73 to 4.19]
  Change at Cycle 10: number analyzed (Participants) | 148 | 163 | 163
  Change at Cycle 10 | 1.52 [-0.96 to 4] | 1.56 [-0.88 to 3.99] | 1.62 [-0.89 to 4.12]
  Change at Cycle 11: number analyzed (Participants) | 99 | 115 | 110
  Change at Cycle 11 | 0.35 [-2.29 to 3] | 2.72 [0.15 to 5.3] | 2.19 [-0.46 to 4.84]
  Change at Cycle 12: number analyzed (Participants) | 82 | 97 | 98
  Change at Cycle 12 | 1.04 [-1.7 to 3.79] | 3.08 [0.43 to 5.73] | 0.75 [-1.95 to 3.46]
  Change at Cycle 13: number analyzed (Participants) | 57 | 85 | 81
  Change at Cycle 13 | 2.13 [-0.85 to 5.11] | 1.78 [-0.94 to 4.5] | 0.82 [-1.98 to 3.62]
  Change at Cycle 14: number analyzed (Participants) | 54 | 78 | 71
  Change at Cycle 14 | -0.13 [-3.15 to 2.89] | 1.59 [-1.18 to 4.36] | -0.07 [-2.95 to 2.81]
  Change at Cycle 15: number analyzed (Participants) | 44 | 71 | 63
  Change at Cycle 15 | -2.1 [-5.29 to 1.09] | 1.29 [-1.53 to 4.11] | 1.49 [-1.47 to 4.45]
  Change at Cycle 16: number analyzed (Participants) | 42 | 58 | 57
  Change at Cycle 16 | -2.26 [-5.49 to 0.97] | 1.23 [-1.73 to 4.19] | 1.44 [-1.59 to 4.47]
  Change at Follow-up 1: number analyzed (Participants) | 173 | 183 | 171
  Change at Follow-up 1 | -0.96 [-3.38 to 1.47] | -1.26 [-3.66 to 1.14] | -1.62 [-4.11 to 0.86]
  Change at Follow-up 2: number analyzed (Participants) | 143 | 127 | 132
  Change at Follow-up 2 | -0.07 [-2.56 to 2.42] | -1.12 [-3.65 to 1.41] | -1.05 [-3.62 to 1.53]
  Change at Follow-up 3: number analyzed (Participants) | 109 | 101 | 99
  Change at Follow-up 3 | -0.32 [-2.92 to 2.28] | -1.67 [-4.29 to 0.96] | -1.98 [-4.68 to 0.72]
  Change at Follow-up 4: number analyzed (Participants) | 87 | 71 | 81
  Change at Follow-up 4 | -0.91 [-3.62 to 1.8] | -2.54 [-5.36 to 0.29] | -1.03 [-3.84 to 1.78]
  Change at Follow-up 5: number analyzed (Participants) | 70 | 62 | 76
  Change at Follow-up 5 | -2.15 [-4.99 to 0.69] | -5.36 [-8.27 to -2.44] | -0.82 [-3.67 to 2.02]
  Change at Follow-up 6: number analyzed (Participants) | 58 | 45 | 55
  Change at Follow-up 6 | -1.77 [-4.75 to 1.2] | -5.32 [-8.49 to -2.16] | -2.76 [-5.82 to 0.3]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (up to 83 months) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first dose of study drug until 30 days after the last administration of study drug). Analysis was performed on safety population, which was randomized participants who received study drug and analyzed according to the treatment actually received.
Arm/Group | Docetaxel 75 mg/m^2 | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Serious Adverse Events (participants affected / at risk) | 126/387 | 127/369 | 188/391
Other Adverse Events (participants affected / at risk) | 353/387 | 323/369 | 354/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 75 mg/m^2 (N=387) | Cabazitaxel 20 mg/m^2 (N=369) | Cabazitaxel 25 mg/m^2 (N=391)
Abscess intestinal (Infections and infestations) | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 2 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 3
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 5 | 1 | 3
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 12 | 3 | 21
Neutropenic sepsis (Infections and infestations) | 3 | 1 | 4
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 3 | 12
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 | 3
Septic shock (Infections and infestations) | 1 | 0 | 3
Skin infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 9 | 8
Urosepsis (Infections and infestations) | 0 | 1 | 2
Wound infection (Infections and infestations) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 8 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 27 | 7 | 40
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 10
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 5
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 2
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2
Coma (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 3 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 4 | 0
Syncope (Nervous system disorders) | 1 | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 3 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Cataract subcapsular (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 4
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 2 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 9
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 4
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 10
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 2
Necrotising colitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1
Cystitis glandularis (Renal and urinary disorders) | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 10 | 13
Hydronephrosis (Renal and urinary disorders) | 1 | 5 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 2
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder rupture (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 3 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 6 | 3
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 4 | 2
Fatigue (General disorders) | 2 | 2 | 0
General physical health deterioration (General disorders) | 1 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 4
Sudden cardiac death (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 3
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device issue (Product Issues) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 75 mg/m^2 (N=387) | Cabazitaxel 20 mg/m^2 (N=369) | Cabazitaxel 25 mg/m^2 (N=391)
Nasopharyngitis (Infections and infestations) | 25 | 19 | 15
Urinary tract infection (Infections and infestations) | 7 | 35 | 33
Neutropenia (Blood and lymphatic system disorders) | 8 | 11 | 25
Decreased appetite (Metabolism and nutrition disorders) | 66 | 50 | 74
Insomnia (Psychiatric disorders) | 28 | 24 | 20
Dizziness (Nervous system disorders) | 25 | 27 | 34
Dysgeusia (Nervous system disorders) | 70 | 41 | 59
Headache (Nervous system disorders) | 31 | 21 | 27
Paraesthesia (Nervous system disorders) | 24 | 25 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 97 | 43 | 48
Lacrimation increased (Eye disorders) | 37 | 8 | 3
Hypertension (Vascular disorders) | 16 | 20 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 26 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 36 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 10 | 17
Abdominal pain (Gastrointestinal disorders) | 14 | 34 | 33
Constipation (Gastrointestinal disorders) | 69 | 90 | 78
Diarrhoea (Gastrointestinal disorders) | 140 | 120 | 190
Dyspepsia (Gastrointestinal disorders) | 13 | 20 | 15
Nausea (Gastrointestinal disorders) | 86 | 92 | 125
Stomatitis (Gastrointestinal disorders) | 53 | 18 | 26
Vomiting (Gastrointestinal disorders) | 44 | 44 | 75
Alopecia (Skin and subcutaneous tissue disorders) | 151 | 33 | 51
Nail disorder (Skin and subcutaneous tissue disorders) | 35 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 23 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 34 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 52 | 64 | 55
Bone pain (Musculoskeletal and connective tissue disorders) | 24 | 31 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 28 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 22 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 | 26 | 19
Dysuria (Renal and urinary disorders) | 9 | 23 | 21
Haematuria (Renal and urinary disorders) | 13 | 69 | 91
Asthenia (General disorders) | 94 | 84 | 90
Fatigue (General disorders) | 110 | 105 | 126
Oedema peripheral (General disorders) | 78 | 36 | 30
Pyrexia (General disorders) | 36 | 22 | 28
Blood creatinine increased (Investigations) | 14 | 27 | 16
Weight decreased (Investigations) | 19 | 17 | 40
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 6 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.